CLINICAL TRIAL: NCT04561804
Title: NAFLD and Liver Fibrosis in Obese Adolescents Undergoing Weight Loss by Surgery or Life Style Intervention
Brief Title: NAFLD and Liver Fibrosis in Obese Adolescents
Acronym: NAFLD
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Prof Shlomi Cohen, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0097-17-TLV
Record Dates: First submitted 2020-09-17; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Liver Fibrosis; Liver Steatosis; Weight Loss
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver; Weight Loss | interventions — Diet Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LISESTYLE INTERVENTION: LOW CARB LOW GLYCEMIC LOAS DIET
- WEGHT LOSS SURGERY: SLEEVE OR MINBYPASS SURGERY
  Interventions: Procedure: laparoscopic sleeve gastrectomy (LSG) and laparoscopic single anastomosis gastric bypass (LSAGB)

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy (LSG) and laparoscopic single anastomosis gastric bypass (LSAGB) — The participants will receive nutritional recommendations for a low carbohydrate, low glycemic load, and isocaloric diet. The diet will be composed of carbohydrates (CHO;35%), fats (40-50%), and proteins (20-25%), and will be tailored to individual preferences and calorie requirements. The number of CHO, protein and fat servings will be determined based on the recommended total energy requirements for age, calculated on the basis of dietary reference intake (DRI). Participants will not be instructed to restrict calories, but to reduce carbohydrate based on their glycemic load.
  The subjects will be instructed about appropriate food choices, and each subject was provided a diet information booklet containing food list, sample menus and recipes
  Other Names: Dietary intervention
  Groups: WEGHT LOSS SURGERY

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a chronic liver disease resulting from excessive fat accumulation in the liver. Due to its close association with obesity, it has become the most common liver disease in children in the United States. NAFLD can result in progressive fibrosis and lead to end-stage liver disease. Best practices in management of pediatric NAFLD are not clearly defined.

Our aim is to clarify the natural history of NAFLD in obese children after weight loss surgery compare to lifestyle intervention. Our secondary aim is to investigate the added value of elastography for the screening and diagnosis of NASH with fibrosis.

DETAILED DESCRIPTION:
The study population will consist of obese adolescents, male and female, age 7-18, that will go through weight loss reduction surgery (WLS) in the Obesity Clinic at Tel Aviv Sourasky Medical Center. A control group matched for age and sex will consist of patients that will go through conventional treatment (see below) at the Obesity Clinic in Dana Dwek Children's Hospital.

Written informed consent form will be signed by the participant before enrollment Patient Population Patients with a diagnosed primary liver disease (autoimmune liver disease, metabolic liver disease, Wilson's disease, alpha 1 antitrypsin deficiency), patients treated with medications known to induce steatosis (such as valproate, amiodarone or prednisone), and patients with hepatic virus infections or history of parenteral nutrition were excluded from the study.

Study Design and measurements This clinical trial aims to asses the effect of bariatric surgery and dietary intervention on hepatic fibrosis in obese pediatric population with NAFLD (Clinical Trial Registration- MOH_2017-06-07_000470, https://my.health.gov.il/CliniTrials/Pages/MOH_2017-06-07_000470.aspx). At the initial visit, data were collected on socioeconomic parameters, lifestyle, birth details, and medical, family, and social histories. All patients underwent anthropometric measures (height, weight and BMI) and a physical examination focused on obesity-related conditions. Laboratory evaluation included liver enzyme profile, lipid profile, glucose, insulin, and HbA1C. Liver fibrosis was estimated by Shearwave elastography (Supersonic) and categorized into 4 levels, F0-F4, according to liver stiffness (measured by kPa), as recently demonstrated elsewhere [9]. Liver steatosis was calculated by a hepatorenal index (HRI) and divided into 3 levels of severity. All measurements were taken by a single experienced radiologist (MW), who was blinded to the results of other parameters of the patients. A multidisciplinary team included a gastroenterologist, hepatologists, a registered dietitian (RD) and a psychologist. All participants received nutritional recommendations (see below) and general recommendation for a healthy lifestyle (regular engagement in daily physical activity and reduction of screen time). Compliance with the dietary guideline was reviewed by a RD on a biweekly basis with a 3-day food questionnaire (2 weekdays and 1 day of the weekend). Blood tests and elastography were repeated after 3 months of intervention.

Determination of the BMI percentiles for age and gender was based on WHO growth charts. "Obesity" was defined as a BMI >95th percentile . Abnormal glucose metabolism included taking a hypoglycemic medication or having an elevated homeostatic model assessment index of insulin resistance, glucose, or HBA1c. Hypertriglyceridemia and hypercholesterolemia were defined as a serum level >95 percentile for age and sex. Hypertension was diagnosed as systolic and/or diastolic blood pressure ≥95 percentile for age and sex. Patients with clinical suspicion of obstructive sleep apnea (OSA) were diagnosed by polysomnography that was conducted by the hospital's sleep specialists. Socioeconomic status was defined according to parents' years of education.

The dietary intervention The participants received nutritional recommendations for a low carbohydrate, low glycemic load, and isocaloric diet. The diet was composed of carbohydrates (CHO;30-40%), fats (35-50%), and proteins (20-25%), and was tailored to individual preferences and calorie requirements. The number of CHO, protein and fat servings was determined based on the recommended total energy requirements for age, calculated on the basis of dietary reference intake (DRI). Participants were not instructed to restrict calories, but to reduce carbohydrate based on their glycemic load. High glycemic index (GI) carbohydrate intake (refined grains, potatoes, sweet and salted snacks and sugar sweetened beverages) was completely restricted, low GI carbohydrates (non-starchy vegetables, legumes, nuts,) were allowed and some low /moderate GI carbohydrate were allowed but limited such as fruits and whole grain bread.

The subjects were instructed about appropriate food choices, and each participant was provided a diet information booklet containing food list, sample menus and recipes

Statistical Analyses Descriptive statistics were examined for all variables. Continuous variables were expressed as median with interquartile range (IQR) when they were not normally distributed and as mean ± standard deviation (SD) for normally distributed variables. Categorical variables were presented as number and percentage. Categorical variables were compared by the McNamer test and continuous and ordinal variables by the Wilcoxon test. The Fischer test was used when the McNamer test was not applicable for some variables. The Pearson correlation and simple linear regression analysis were performed to examine bivariate associations between fibrosis and metabolic and nutritional parameters. The Wilcoxon signed rank test was applied to compare the difference between steatosis, fibrosis, and metabolic parameters between the 2 time points (baseline and 3-month follow-up). A P level <0.05 was considered statistically significant. All statistical tests were 2-sided. The statistical analysis was performed with SPSS (IBM SPSS statistics, version 22, IBM Corp. Armonk, NY, USA, 2013.).

ELIGIBILITY:
IInclusion criteria:

* Age 13-18 years.
* No other chronic disease except the metabolic syndrome.
* Not taking any medication

Exclusion criteria:

* Children that are known to suffer from genetic/metabolic disorders that can cause steatosis- Wilson disease, hypothyroidism, autoimmune hepatitis, Alpha 1 antitrypsin.
* Children infected with HBV or HCV, HAV.
* Children that use medications that can cause liver steatosis- amiodarone, MTX, Corticosteroids
* Children with significant ethanol consumption ->10 gr per day for women and >20gr per day for men.
* Pregnant women.
* Obesity due to syndromes or monogenic disease

General withdraw criteria:

• If the participant withdraws his consent.

Age Groups: Child, Adult, Older Adult
Study Population: We prospectively recruited all children and adolescents (age 7-18 years) with obesity who were admitted to the Obesity clinic at Dana-Dwek Children's Hospital of the Tel Aviv Medical Center between December 1, 2018, and December 1, 2019. All children with a BMI >95 percentile for age were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
change in liver fibrosis | 3 and 6 months
  Liver fibrosis will be estimated by Shearwave elastography (Supersonic) and categorized into 4 levels, F0-F4, according to liver stiffness

SECONDARY OUTCOMES:
change in liver steatosis | 3 and 6 months
  Liver steatosis will be calculated by a hepatorenal index (HRI) and divided into 3 levels of severity
weight reduction | 3 and 6 months
  BMI measurements

CONTACTS AND LOCATIONS:
Overall Officials: sHLOMI Cohen, prof, Principal Investigator — Dana Dwek Children Hospital
Locations (1):
- Pediatric Gastroenterology, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
The data will be provided to other researchers upon a reasonable request

REFERENCES:
- [Derived] Moran-Lev H, Cohen S, Webb M, Yerushalmy-Feler A, Amir A, Gal DL, Lubetzky R. Higher BMI predicts liver fibrosis among obese children and adolescents with NAFLD - an interventional pilot study. BMC Pediatr. 2021 Sep 3;21(1):385. doi: 10.1186/s12887-021-02839-1. PMID 34479517
- Available data/document: Study Protocol — https://my.health.gov.il/CliniTrials/Pages/MOH_2017-06-07_000470.aspx — Israel Ministry of Health registration number